CLINICAL TRIAL: NCT01326624
Title: Study of the Wearable Defibrillator In Heart-Failure Patients
Acronym: SWIFT
Status: Completed | Type: Observational
Sponsor: Zoll Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 90D0112
Record Dates: First submitted 2011-03-29; First posted 2011-03-31 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Heart Failure; Ventricular Dysfunction; Sudden Death; Sudden Cardiac Arrest; Ventricular Tachycardia; Ventricular Fibrillation
Keywords: heart failure; ventricular dysfunction; sudden death; sudden cardiac arrest; ventricular tachycardia; ventricular fibrillation; wearable defibrillator
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction; Death, Sudden; Death, Sudden, Cardiac; Tachycardia, Ventricular; Ventricular Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- NYHA class III or IV: Patients with NYHA class III or IV during the past month and one or more of the following:
  * Hospitalization for cardiac decongestion and stabilization.
  * Advanced heart failure receiving intravenous diuretics/inotropics in an outpatient clinic.
  * Awaiting cardiac transplantation
  Interventions: Device: wearable defibrillator (LifeVest)
- left ventricular ejection fraction ≤ 35%: Patients with left ventricular ejection fraction ≤ 35% and either one of the following:
  * Coronary revascularization within 3 calendar months prior to enrollment.
  * Heart failure of non-ischemic origin diagnosed within 3 calendar months prior to enrollment.
  Interventions: Device: wearable defibrillator (LifeVest)
- Awaiting ICD re-implantation
  Interventions: Device: wearable defibrillator (LifeVest)
- Acute myocardial infarction: Patients hospitalized with acute myocardial infarction and Killip Class III/IV.
  Interventions: Device: wearable defibrillator (LifeVest)

INTERVENTIONS:
Device: wearable defibrillator (LifeVest) — LifeVest wearable defibrillator for unattended treatment of sudden cardiac arrest due to ventricular tachycardia or ventricular fibrillation
  Other Names: wearable cardioveter defibrillator; WCD; LifeVest

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of wearable defibrillator use in patients with left ventricular dysfunction or advanced heart failure symptoms, who have a high-risk for sudden cardiac death but are either not eligible for an implantable defibrillator under current guidelines or are not able to receive the device due to their condition.

ELIGIBILITY:
Inclusion Criteria:

* Patients with NYHA class III or IV during the past month and one or more of the following:

  * hospitalization for cardiac decongestion and stabilization,
  * advanced heart failure receiving intravenous diuretics/inotropics in an outpatient clinic, or
  * awaiting cardiac transplantation
* Patients with left ventricular ejection fraction ≤ 35% and either one of the following:

  * coronary revascularization within 3 calendar months prior to enrollment, or
  * heart failure of non-ischemic origin diagnosed within 3 calendar months prior to enrollment.
* Patients awaiting ICD re-implantation following device explantation or lead extraction,
* Patients hospitalized with acute myocardial infarction and Killip Class III/IV.

Exclusion Criteria:

* The presence of an implantable cardioverter defibrillator prior to enrollment.
* Advanced cerebrovascular disease.
* Non-cardiac terminal illness associated with reduced likelihood of survival for the duration of the study.
* Use of supplemental oxygen in an outpatient setting requiring an external oxygen tank.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with left ventricular dysfunction or advanced heart failure symptoms (New York Heart Association functional Class III/IV), who have a high-risk for sudden cardiac death, but are not eligible for an implantable defibrillator or are not able to receive one due to their condition.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2011-03; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Defibrillation for life-threatening ventricular tachyarrhythmias | 6 months
Assess magnitude and complexity of ventricular and atrial arrhythmias during use | 6 months

SECONDARY OUTCOMES:
Total mortality | 6 months and 12 months
Compliance with wearable defibrillator use | 6 months
Quality of life with a wearable defibrillator | 6 months
Complications (adverse events) with wearable defibrillator use | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Eldar, MD, Principal Investigator — Chaim Sheba Medical Center
Locations (2):
- University of Rochester, Rochester, New York, United States
- Chaim Sheba Medical Center, Tel Litwinsky, Israel